CLINICAL TRIAL: NCT03238404
Title: The Application of Neoadjuvant Chemotherapy for Patients With Advanced Gastric Cancer in Enhanced Recovery After Surgery Programs for Radical Gastrectomy
Brief Title: Neoadjuvant Chemotherapy for Patients With Advanced Gastric Cancer in ERAS Programs for Radical Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JIANG Zhi-Wei (Other)
Responsible Party: Sponsor-Investigator, JIANG Zhi-Wei, Vice director of Research Institute of General Surgery, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BE2015687NAC
Record Dates: First submitted 2017-07-27; First posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; neoadjuvant chemotherapy; enhanced recovery after surgery; gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a single-center, parallel, open-label randomized controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAC group (Experimental): Patients will receive neoadjuvant chemotherapy (NAC) before the gastrectomy and ERAS.
  Interventions: Procedure: NAC group
- Surgery alone group (Active Comparator): Patients will not receive NAC before the gastrectomy and ERAS.
  Interventions: Procedure: Surgery alone group

INTERVENTIONS:
Procedure: NAC group — NAC is the name of a procedure. NAC doesn't mean different interventions are used. Patients in this group need receive this NAC procedure instead of one drug before the gastrectomy and ERAS. The program consists of an intravenous injection of 130 mg/m2 oxaliplatin on day 1, followed by oral administration of 50 mg tegafur gimerac (the name of an anticarcinogen) twice daily on days 1-14, every 3 weeks.
  Arms: NAC group
Procedure: Surgery alone group — Patients will not receive neoadjuvant chemotherapy and they will undergo the gastrectomy and ERAS alone.
  Arms: Surgery alone group

SUMMARY:
Patients with advanced gastric cancer received neoadjuvant chemotherapy undergo enhanced recovery after surgery (ERAS) programs.

DETAILED DESCRIPTION:
In recent years, enhanced recovery after surgery (ERAS) programs were applied in gastrectomy in areas with a high prevalence of gastric cancer, such as China and Japan, confirming that ERAS programs accelerate the postoperative rehabilitation of gastric cancer patients without increasing the occurrence rate of postoperative complications. However, in most studies on ERAS for gastric cancer, patients who received neoadjuvant chemotherapy were excluded. Investigators designed this study aimed to evaluate whether patients who receive neoadjuvant chemotherapy can enrolled into enhanced recovery after surgery programs for locally advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with locally advanced gastric cancer.
2. Age older than 18 and younger than 75 years.
3. American Society of Anesthesiologists (ASA) class: I-III.
4. Participants can describe the symptom objectively and cooperate actively.
5. Written informed consent

Exclusion Criteria:

1. Patients allergic to oxaliplatin, tegafur gimerac etc.
2. Patients with ischemic heart disease, cerebrovascular disease and peripheral vascular disease, or cardiac function > II (NYHA)
3. Patients with complications (bleeding, perforation and obstruction) caused by gastric cancer.
4. Patients with severe liver and renal dysfunction (Child - Pugh ≥ 10; Cr < 25 ml/min).
5. Patients who require simultaneous surgery for other diseases.
6. Patients who received upper abdominal surgery previously.
7. Pregnant or breast-feeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-08-10 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
Postoperative length of stay | 1 month
  Postoperative length of stay

SECONDARY OUTCOMES:
Postoperative complications | 2 months
  Postoperative complications
The time to first flatus | 1 week
  Bowel recovery
Time to semi-liquid diet | 2 weeks
  Bowel recovery
Total protein | 1 week
  Nutritional status
Albumin | 1 week
  Nutritional status
Prealbumin | 1 week
  Nutritional status

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Wei JIANG, Ph.D., Principal Investigator — Jinling Hospital, Medical School of Nanjing University; Jian ZHAO, Ph.D., Study Director — Jinling Hospital, Medical School of Nanjing University
Locations (1):
- Jinling Hospital, Medical School of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
The results and IPD will be considered to share in published articles.